CLINICAL TRIAL: NCT02917876
Title: Predictors of De-novo Development of Obstructive Sleep Apnea in Pregnancy
Acronym: Predictors
Status: Active, not recruiting | Type: Observational
Sponsor: The Miriam Hospital (Other)
Collaborators: Brown University (Other); Rhode Island Hospital (Other); Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Ghada Bourjeily, Associate Professor of Medicine, The Miriam Hospital
Other Study IDs: 1R01HL130702 (NIH)
Record Dates: First submitted 2016-09-21; First posted 2016-09-28 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Sleep Apnea; Pregnancy; Obesity; Sleep
Keywords: Obstructive Sleep Apnea; Pregnancy; Obesity; Fluid shifts; Body composition; Sleep
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be stored for future testing
Oversight: Data Monitoring Committee: No

SUMMARY:
This study seeks to understand the physical, physiologic and biologic features that predispose a woman to the development of obstructive sleep apnea once they are exposed to the cardiopulmonary and metabolic physiological changes of pregnancy. Knowing these specific predictive factors can help identify a population at risk and guide clinicians to develop suitable targeting screening strategies.

DETAILED DESCRIPTION:
Patients will be recruited from multiple community and hospital-based practices that care for pregnant women. Subjects will have:

1. measurements of body composition
2. anthropometric measures
3. sleep and mood questionnaires
4. Home sleep studies
5. blood testing for biological markers
6. salivary testing for hormonal markers
7. pulmonary function tests and upper airway patency measurements

Women without sleep apnea at enrollment will then be followed longitudinally for the development of obstructive sleep apnea during pregnancy with repeat assessment during their third trimester. Women diagnosed with sleep apnea at enrollment will have no further assessment in late pregnancy.

Monetary incentives will also be issued at data collection points. Subjects will receive small gift incentives such as baby-related items.

ELIGIBILITY:
Inclusion Criteria:

* <13 completed weeks of gestation
* BMI >30 kg/m2 at recruitment
* >18 years of age
* Ability to give informed consent

Exclusion Criteria:

* Unable to meet inclusion criteria
* Twin pregnancies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women, 18 years or older, at less than 13 completed weeks of gestation and who have a BMI that is greater than 30 kg/m2 at recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2016-11; Primary Completion 2023-12-30 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Characteristics of participants who develop obstructive sleep apnea defined as an apnea hypopnea index >5 events per hour | Up to 40 weeks
  The study will develop a model of biologic, physiologic and anthropometric measures that predict the development of obstructive sleep apnea apnea later in pregnancy compared to baseline in early pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Bourjeily, MD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available within 12 months of study completion.
Access Criteria: Investigators data access requests will be reviewed by an independent review committee. Requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Bublitz MH, Nillni Y, Nugent NR, Sanapo L, Habr N, Bourjeily G. Posttraumatic stress disorder, diurnal cortisol, and ambulatory blood pressure in early and late pregnancy. J Trauma Stress. 2023 Feb;36(1):239-246. doi: 10.1002/jts.22895. Epub 2022 Dec 4. PMID 36464928
- [Derived] Sanapo L, Bublitz MH, Bai A, Mehta N, Messerlian GM, Catalano P, Bourjeily G. Association between sleep disordered breathing in early pregnancy and glucose metabolism. Sleep. 2022 Apr 11;45(4):zsab281. doi: 10.1093/sleep/zsab281. PMID 34999843